CLINICAL TRIAL: NCT06720844
Title: Idiopathic Central Precocious Puberty and Associated Neurodevelopmental Syndromes and Pathologies: Evaluation of Frequency and Comparison of Diagnostic and Developmental Characteristics
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SDR-PPC23
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Central Precocious Puberty (CPP)
Keywords: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Observational, retrosopective, single-centre, non-profit study focused on the frequency of Central Precocious Puberty idiopathic, or associated to Neurodevelopmental Syndromes and Pathologies, and comparison of diagnostic and developmental characteristics of patients.

DETAILED DESCRIPTION:
The study enrolls both male and female patients referred to the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria Policlinico di Sant'Orsola between 01/01/2013 and 31/12/2023 for Central Precocious Puberty and treated with GnRH analouge. The primary aim of the study is to Assess the frequency of diagnosis of idiopathic or syndromic Central Precocious Puberty in the last decade. The secondary aims are to Compare clinical, laboratory and instrumental characteristics at diagnosis and in follow-up between patients with idiopathic and syndromic PPC, and to identifying possible pathogenetic factors characterising different forms of Central Precocious Puberty.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Central Precocious Puberty presenting an indication to undertake treatment with GnRH analogue: Appearance of secondary sexual characteristics (thelarche or gonadarche) before the age of 8 for females and 9 for males; Acceleration of the rate of statural growth and advancement of bone age one year older than the chronological age; LH peak > 5 IU/L on GnRH test and a longitudinal uterine diameter > 36 mm in females, with or without the appearance of endometrial rhyme;
* Age at onset of entral Precocious Puberty between 2 and 8 years (females) or between 2 and 9 years (males);
* Age at enrollment < 18 years;
* Follow-up of at least 12 months;
* Obtaining informed consent from parents/legal guardian of peduatric patients.

Exclusion Criteria:

* Isolated telarche and/or pubarche;
* Peripheral forms of precocious puberty;
* Patients diagnosed with primary organic Central Precocious Puberty due to tumour- or non-tumour-causing hypothalamic lesions.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All male and female patients referred to the Pediatrics Unit of the IRCCS Azienda Ospedaliero-Universitaria Policlinico di Sant'Orsola between 01/01/2013 and 31/12/2023 for Central Precocious Puberty and treated with GnRH analouge.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-03-13 (Estimated); Study Completion 2025-05-13 (Estimated)

PRIMARY OUTCOMES:
Frequency of diagnosis of idiopathic or syndromic Central Precocious Puberty | at baseline
  diagnosis of idiopathic or syndromic Central Precocious Puberty

CONTACTS AND LOCATIONS:
Overall Officials: Federico Baronio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bolgona, Italy